CLINICAL TRIAL: NCT03981328
Title: The Effectiveness of Real Time Continuous Glucose Monitoring to Improve Glycemic Control and Pregnancy Outcome in Patients With Gestational Diabetes Mellitus
Brief Title: Real-time Continuous Glucose Monitoring for Reduced Adverse Complications and Events in Women With Gestational Diabetes (GRACE): a Multicentre International Randomized Controlled Trial
Acronym: GRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Charite University, Berlin, Germany (Other); CNR Institute of Neurosceince, Padova, Italy (Unknown); Università Politecnica delle Marche (Other); DexCom, Inc. (Industry); Jena University Hospital (Other); German Diabetes Center (Other)
Responsible Party: Principal Investigator, Christian Göbl, Principal Investigator, Privatdozent, MD, PhD, MSc, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20181101
Record Dates: First submitted 2019-02-15; First posted 2019-06-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cgm; Gestational Diabetes; Pregnancy Complications; Blood Glucose; GDM
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- self-monitored blood glucose (Active Comparator): The control group participants will perform self-monitored blood glucose testing with a study-provided blood glucose meter, including testing supplies. They will perform capillary blood glucose monitoring as routinely used for patients with GDM i.e. at least four capillary blood glucose values daily including measurements at fasting as well as 1h after starting each meal by using a routinely available blood glucose measurement device.
  Interventions: Device: self-monitored blood glucose
- Continuous glucose monitoring (Experimental): Patients randomized to the intervention group will be equipped with a real-time CGM sensor (Dexcom G6 sensor, a small flexible device that records interstitial glucose levels every five minutes). The sensor will be inserted into the subcutaneous tissue of the anterior abdomen wall. Additionally, patients will be advised to record capillary blood glucose values if glucose alerts or readings do not match with symptoms or expectations. Participants will be educated how to exchange the sensor (has to be exchanged every ten days) and will be equipped with a real-time CGM monitor and instructed in its use. The monitor provides the user with information about current glucose levels and notifies the patient before she reaches her upper or lower glucose threshold and when glucose levels change rapidly. All patients in the intervention group will specifically trained how to use the system.
  Interventions: Device: Dexcom G6 Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Dexcom G6 Continuous Glucose Monitoring System — Users insert a tiny sensor wire just under their skin using an automatic applicator. The sensor can measure glucose readings in interstitial fluid throughout the day and night.
  Arms: Continuous glucose monitoring
Device: self-monitored blood glucose — Each participant in the control group will be assigned a study blood glucose meter to measure and store their blood glucose values during the study. Therefore, the Contour® Next One system (or a comparable device) will be used. The meter has CE Mark clearance and is commercially available in Europe. Participants will receive an ample supply of meter test materials based on quantities routinely used.
  Arms: self-monitored blood glucose

SUMMARY:
Real-time continuous glucose monitoring (CGM) systems provide users with information about current glucose levels and alert the patient before the upper or lower glucose threshold is reached or when glucose levels change rapidly. Hence, glycaemic excursions can be early identified and accordingly adapted by behavioural change or pharmacologic intervention. Randomized controlled studies adequately powered to evaluate the impact of long-term application of real-time CGM systems on the risk reduction of adverse obstetric outcomes are missing.

DETAILED DESCRIPTION:
Intervention: Device description The Dexcom G6 intended use is for the management of diabetes in persons aged 2 years and older. The Dexcom G6 System is intended to replace fingerstick blood glucose testing for diabetes treatment decisions. Interpretation of the Dexcom G6 System results should be based on the glucose trends and several sequential readings over time. The Dexcom G6 System also aids in the detection of episodes of hyperglycemia and hypoglycemia, facilitating both acute and long-term therapy adjustments. The Dexcom G6 System can be used alone or in conjunction with these digitally connected medical devices for the purpose of managing diabetes. The system consists of a sensor, transmitter, receiver, and mobile app. The sensor is a small, flexible wire inserted into subcutaneous tissue where it converts glucose into electrical current. The sensor incorporates an interferent layer that minimizes the effect of potential electroactive interferents, such as acetaminophen, by preventing it from reaching the sensor wire surface. The benefit of this interferent layer in blocking the effects of acetaminophen prevents falsely high glucose readings. Thus, users may ingest acetaminophen while wearing the G6 CGM system. The transmitter, which is connected to the sensor and worn on the body, samples the electrical current produced by the sensor and converts the measurement into a glucose reading using an onboard algorithm. The receiver and/or the app displays the glucose reading along with a rate of change arrow and a trend graph. Additionally, the receiver and/or app issues alarms and alerts to notify the patient of glucose level changes and other important system conditions. The app provides the additional capability to share data with "followers" using the Dexcom Share service. The receiver can be put into a blinded mode using CLARITY® software. In this mode, users are unable to see the CGM data or receive CGM alerts.

CGM Ancillary Devices Dexcom CLARITY® is an accessory to users of the Dexcom CGM system. It is a software program that allows the transfer of glucose data from the CGM system to Dexcom remote servers for data management to allow use of the CGM data by the user and study clinicians. Target ranges of 60 to 140 mg/dl [3.3 to 7.8 mmol/l] will be set and the patients will be introduced in the use of alarm settings. Both participants and study sites will use CLARITY® to transfer glucose data between user and study site, whether CGM is used in blinded or real-time mode. A CLARITY® mobile app can be used for retrospective review of glucose data on the smart device and can also be set up to allow receipt of push notifications of CGM data facilitating weekly data review. For all patients (intervention and control group) an anonymized CLARITY® account will be created by using a sequential study number which is allocated at randomization (sex will be female and birth date for each account will be set to 1.1.1990 for all accounts).

1. For participants that have a supported phone, the G6 CGM app will be installed on participant's smart phone.
2. An anonymized CLARITY® mobile account will be set up and linked to the research site.
3. Participants will use CGM data for their diabetes management.

5. A high alert threshold will be set at 140 mg/dl [7.8 mmol/l]. Low alert threshold and urgent low soon alerts will be turned off. If participants require insulin, the low alert will be turned on and the threshold set at 65 mg/dl [3.6 mmol/l]. In addition, the urgent low alert (55 mg/dl [3.1 mmol/l]), the urgent low soon alert (when glucose levels are falling fast and will be below 55 mg/dl [3.1 mmol/l] in less than 20 min) as well as alerts for rise and fall rate (3 mg/dl [0.17 mmol/l]) in addition to alerts for signal loss and no readings for more than 20 min will be enabled. 6. Participants with applicable smart phones may have CLARITY® push notifications on the CLARITY® mobile app about weekly time in range comparison enabled during the study.

7. For app users, the "Share and Follow" functionality will be discussed and encouraged (i.e.

the study participants are able to invite followers to review their glucose levels).

8. For participants using the receiver only, the receiver will be downloaded into the CLARITY® clinic account at each visit. 9. For participants using real-time CGM data summary will be downloaded for documentation at V3 and V4 (between 36+0 and 38+6) as well as after delivery (VPP1) 10. The research team will review the CGM in CLARITY® to inform lifestyle and therapy recommendations. 11. The Dexcom G6 system will not be calibrated during the study period.

ELIGIBILITY:
Inclusion Criteria:

* female patients between 18 and 55 years
* gestational diabetes mellitus in accordance with the IADPSG criteria between 24 and 31+6 weeks of gestation by a 2h 75g OGTT
* If the GDM diagnosis is made before 24+0 weeks of gestation in accordance with the local guideline (i.e. when IADPSG cut-offs for fasting and post-load glucose are exceeded) patients can be included if no insulin treatment was started until 24+0

Exclusion Criteria:

* Overt diabetes (i.e. pregestationally known type 1 or type 2 diabetes or fasting plasma glucose during the OGTT ≥126 mg/dl [7.0 mmol/l] or HbA1c ≥6.5% [44 mmol/l] or 2h post-load OGTT levels ≥200 mg/dl [11.1 mmol/l] assessed before 24+0 weeks of gestation
* history of bariatric surgery or other surgeries that induce malabsorption
* long-term use (>2 weeks) of systemic steroids prior to enrolment
* multiple pregnancy
* Patients already using glucose lowering medications (metformin or insulin) before study entry
* fetal growth restriction due to placental dysfunction at study entry - Inpatient psychiatric treatment up to 1 year before enrolment
* Participation in this study in previous pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 375 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
LGA newborns | postpartum - up to 48 hours after delivery
  To assess differences in the proportion of LGA newborns (birth weight >90. pct) in women with GDM using real-time CGM as compared to women with GDM using SMBG via capillary blood glucose monitoring.

SECONDARY OUTCOMES:
neonatal hypoglycaemia | postpartum - up to 48 hours after delivery
  newborn measurement
rate of caesarean section | postpartum - up to 48 hours after delivery
  statistics
shoulder dystocia | postpartum - up to 48 hours after delivery
  frequency of occurrences
neonatal anthropometry | postpartum - up to 48 hours after delivery
  newborn measurement
differences in neonatal hyperinsulinemia | postpartum - up to 48 hours after delivery
  differences in neonatal hyperinsulinemia
CGM measures such as mean, glycaemic variability, time in range as well as hyper- and hypoglycaemia | through study completion, an average of 9 months
  maternal measurements
duration and frequency postprandial hyperglycaemic excursions | through study completion, an average of 9 months
  maternal
start and amount of glucose lowering therapy | through study completion, an average of 9 months
  development until birth
HbA1c | through study completion, an average of 9 months
  maternal measurements
glycosylated Fibronectin | through study completion, an average of 9 months
  maternal measurements
change in bodyweight during pregnancy and after delivery as well as glucose disposal at postpartum | through study completion, an average of 1 year
  development until birth
Health-related quality of life | through study completion, an average of 9 months
  development until birth

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Division of Obstetrics and Feto-maternal Medicine, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Linder T, Dressler-Steinbach I, Wegener S, Schellong K, Schmidt S, Eppel D, Monod C, Heinzl F, Redling K, Winzeler B, Mosimann B, Weschenfelder F, Groten T, Mittlbock M, Jendle J, Henrich W, Morettini M, Bozkurt L, Tura A, Gobl C; GRACE study collaborative group. Glycaemic control and pregnancy outcomes with real-time continuous glucose monitoring in gestational diabetes (GRACE): an open-label, multicentre, multinational, randomised controlled trial. Lancet Diabetes Endocrinol. 2026 Jan;14(1):50-61. doi: 10.1016/S2213-8587(25)00288-8. Epub 2025 Nov 24. PMID 41308662
- [Derived] Huhn EA, Linder T, Eppel D, Weisshaupt K, Klapp C, Schellong K, Henrich W, Yerlikaya-Schatten G, Rosicky I, Husslein P, Chalubinski K, Mittlbock M, Rust P, Hoesli I, Winzeler B, Jendle J, Fehm T, Icks A, Vomhof M, Greiner GG, Szendrodi J, Roden M, Tura A, Gobl CS. Effectiveness of real-time continuous glucose monitoring to improve glycaemic control and pregnancy outcome in patients with gestational diabetes mellitus: a study protocol for a randomised controlled trial. BMJ Open. 2020 Nov 30;10(11):e040498. doi: 10.1136/bmjopen-2020-040498. PMID 33257486

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03981328/Prot_SAP_000.pdf